CLINICAL TRIAL: NCT03885765
Title: Complication and Lung Function Impairment Prediction Using Perfusion and CT Air Trapping (CLIPPCAIR): Protocol for the Development and Validation of a Novel Algorithm for Post-resection Lung Function
Brief Title: Complication and Lung Function Impairment Prediction Using Perfusion and CT Air Trapping
Acronym: CLIPPCAIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0370
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 40 resected lung tissues for the routine pathological analysis may be retained for ancillary studies if the investigator :
  * deems that sample recovery is feasible
  * judges the distance between the cancerous lesion and the region of interest, sufficiently large/distinct
  * obtained the patient's consent for the use of his remaining excised tissue specifically for this ancillary study
  These lung tissues can't be retained if :
  * unavailability of tissue sample due to routine analysis requirements
  * patient has atelectasis
  * patient has pulmonary infection
  * patient has a pulmonary lesion linked to the surgical intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: The first 60 patients recruited.
  Interventions: Diagnostic Test: Predictive data; Procedure: Lung resection
- Validation group: The last 100 patients recruited.
  Interventions: Diagnostic Test: Predictive data; Procedure: Lung resection

INTERVENTIONS:
Diagnostic Test: Predictive data — The novel predictive data in this study includes 5 predefined variables derived from thoracic CT scans:
  (i) Expiratory to inspiratory ratio of mean lung density (MLDe/i), total; (ii) MLDe/i of the section to be excised / MLDe/i total; (iii) Percentage of emphysema according to voxel thresholding at -950 HU (PVOX-950), total; (iv) PVOX-950 for the section to be excised; (v) Iodine concentration [I] of the section to be excised / [I] total.
Procedure: Lung resection — Surgical resection will be characterised by type (pneumonectomy, bi-lobectomy, lobectomy, or lobectomy with anastomosis resection), whether or not lymph node dissection was performed, and whether or not the resection was atypical.

SUMMARY:
The primary objective of the CLIPPCAIR study is to construct and validate a new algorithm for predicting post-operative forced expiratory volume in 1 second (FEV1) values for lung resection candidates; this new model will be based on data derived from a thoracic CT scan with injection of contrast media.

DETAILED DESCRIPTION:
Secondarily, the predictions made using traditional scintigraphic data will be compared with those from the new algorithm in a subset of high-risk patients, and cumulative contrast media and irradiation doses associated with imaging will be presented. How other measures of pulmonary function (e.g. transfer factor of the lung for carbon monoxide (TLCO)) and the presence/absence of operative complications might be predicted will also be investigated. Additionally, the potential links between (i) pre-surgical imaging data, (ii) post-surgical changes in respiratory function, and (iii) changes in health related quality of life will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with non-small cell lung cancer
* Indication for pulmonary excision surgery
* Patient requiring a more recent pre-surgical computed tomography scan (CT scan)
* The patient has been correctly informed about the study and has signed the consent form
* The patient is affiliated with or a beneficiary of the French single-payer social security programme (national health insurance)

Exclusion Criteria:

* Patient in an exclusion period determined by another protocol
* Participation in another study that may affect the results of the present study (anti-cancer treatment studies are allowed)
* Patient under legal or judicial protection
* Contraindication to surgery or iodine injection
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted study population corresponds to non-small cell lung cancer patients requiring pulmonary excision and who need to update their computed tomography scan data (CT scan) prior to surgery.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) from spirometry | 6 months
Correlation between predicted and real values for post-surgical FEV1 | 6 months

SECONDARY OUTCOMES:
Estimated post-operative FEV1 (litres) according to scintigraphy | Baseline (day 0)
  Estimated post-operative FEV1 (litres) deduced from the regional FEV1 distribution according to lung scintigraphy
Estimated post-operative TLCO according to scintigraphy | Baseline (day 0)
  estimated post-operative Transfer factor of the lung for carbon monoxide (TLCO) deduced from the regional TLCO distribution
Estimated post-operative FEV1 according segment counting (1) | Baseline (day 0)
  FEV1post-seg-1 = FEV1pre-op x (1 - 0.0526 x N), where N is the number of segments to be excised
Estimated post-operative FEV1 according segment counting (2) | Baseline (day 0)
  FEV1post-seg-2 = FEV1pre-op x [(19 - a - b)/(19 - a)], where a is the number of non-obstructed segments to be excised and b is the number of obstructed segments to be excised
Forced expiratory volume in 1 second (FEV1) from spirometry | Baseline (day 0)
Forced vital capacity from spirometry | Baseline (day 0)
Forced vital capacity from spirometry | 6 months
FEV1/FVC from spirometry | Baseline (day 0)
FEV1/FVC from spirometry | 6 months
Total lung capacity from spirometry | Baseline (day 0)
  lung volumes
Total lung capacity from spirometry | 6 months
  lung volumes
Residual lung volume from spirometry | Baseline (day 0)
  lung volumes
Residual lung volume from spirometry | 6 months
  lung volumes
Functional residual lung capacity from spirometry | Baseline (day 0)
  lung volumes
Functional residual lung capacity from spirometry | 6 months
  lung volumes
Transfer factor of the lung for carbon monoxide (TLCO) from spirometry | Baseline (day 0)
Transfer factor of the lung for carbon monoxide (TLCO) from spirometry | 6 months
Maximum volume of oxygen utilized per unit time (VO2Max) | Baseline (day 0)
Maximum volume of oxygen utilized per unit time (VO2Max) | 6 months
EQ-5D-5L questionnaire | Baseline (day 0)
  The 5 level EQ-5D version (EQ-5D-5L) is a standardized instrument for measuring generic health status. It results in a single index score describing a general health profile ranging from 0 to 1, as well as a visual analogue scale.
EQ-5D-5L questionnaire | 6 months
  The 5 level EQ-5D version (EQ-5D-5L) is a standardized instrument for measuring generic health status. It results in a single index score describing a general health profile ranging from 0 to 1, as well as a visual analogue scale.
QLQ-C30 Version 3.0 questionnaire | Baseline (day 0)
  The QLQ-C30 Version 3.0 (a quality of life questionnaire for lung cancer patients) results in three scale scores [(i) level of function, (ii) global health status, and (iii) symptomatology / problems] with higher scores (ranging from 0 to 100) representing a higher response level.
QLQ-C30 Version 3.0 questionnaire | 6 months
  The QLQ-C30 Version 3.0 (a quality of life questionnaire for lung cancer patients) results in three scale scores [(i) level of function, (ii) global health status, and (iii) symptomatology / problems] with higher scores (ranging from 0 to 100) representing a higher response level.
QLQ-LC13 questionnaire | Baseline (day 0)
  The QLQ-LC13 provide an additional lung-cancer-specific symptom scale ranging from 0 to 100 with higher scores indicating worse symptomatology.
QLQ-LC13 questionnaire | 6 months
  The QLQ-LC13 provide an additional lung-cancer-specific symptom scale ranging from 0 to 100 with higher scores indicating worse symptomatology.
Number of participants with complications | 0 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Bommart, MD, Study Director — University Hospitals of Montpellier, France
Locations (1):
- Chu Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Data will be made available to persons who address a reasonable request to the study director and fulfil the requirements stipulated by the French CNIL (Commission Nationale de l'Informatique et des Libertés : https://www.cnil.fr/professionnel).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Datasets can be requested after the publication process has been completed.
Access Criteria: The conditions under which members of the public will be granted access to datasets are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
  * The appropriate CNIL approval has been obtained by the user.
URL: https://osf.io/2m7z4/

REFERENCES:
- [Background] Suehs CM, Solovei L, Hireche K, Vachier I, Mariano Goulart D, Gamon L, Charriot J, Serre I, Molinari N, Bourdin A, Bommart S. Complication and lung function impairment prediction using perfusion and computed tomography air trapping (CLIPPCAIR): protocol for the development and validation of a novel multivariable model for the prediction of post-resection lung function. Ann Transl Med. 2021 Jul;9(13):1092. doi: 10.21037/atm-21-214. PMID 34423004